CLINICAL TRIAL: NCT04194710
Title: Randomized Clinical Trial Comparing Arthroscopic Debridement Versus Autologous Cytokine Rich Serum for the Treatment of Lateral Epicondylitis
Brief Title: Arthroscopic Debridement Versus Autologous Cytokine Rich Serum for the Treatment of Lateral Epicondylitis
Acronym: DA-SARC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Tecnologia Regenerativa Qrem S.L. (Unknown)
Responsible Party: Principal Investigator, Ferran Fillat Gomà, Co-Investigator, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DA-SARC
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Epicondylitis, Lateral
MeSH Terms: conditions — Tennis Elbow | interventions — Meniscectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthroscopic Resection (Active Comparator): 43 patients will be assigned to this arm. This is the standard technique to treat lateral epicondylitis. After randomization, patients will be informed and the surgery will be scheduled.
  Interventions: Biological: Autologous Cytokine Rich Serum
- Cytokine rich serum injection (Experimental): 43 patients will be assigned to this arm. After randomization, patients will be informed and the first injection of serum rich cytokines will be scheduled. After 15 days, they will be injected again with serum rich cytokines.
  Interventions: Procedure: Arthroscopic Resection

INTERVENTIONS:
Biological: Autologous Cytokine Rich Serum — Proteins, called cytokines, released from blood platelets and leukocytes, play an important role in the repair and regeneration of the injured tissue that causes lateral epicondylitis.
  Autologous Cytokine Rich Serum is prepared by the medical devise Q-Cytokine (CE MED31489) from patient's blood. The company Tecnologia Regenerativa Qrem S.L., with licence number 7096-PS from Agencia Española de Medicamentos y Productos Sanitarios (AEMPS), is the manufacturer of this product. Q-Cytokine is a lab-in-a-box devise, and consist of an automatic centrifuge and a sterile disposable kit. After 9 steps of centrifugation, that take place in 36 minutes, Cytokine Rich Serum is obtained. This Cytokine Rich Serum is then injected to the epicondyle.
  Patients randomized to this treatment will receive 1 injections of Autologous Cytokine Rich Serum right after randomization and another one after 15 days.
  This process will take place at outpatient clinics.
  Arms: Arthroscopic Resection
Procedure: Arthroscopic Resection — Surgical treatment of resection by arthroscopy is the standard treatment for chronic epicondylitis. The surgery is performed in the operating room under local anesthesia and lasts approximately 30 minutes. During the surgery, the doctor accesses the tendon by arthroscopy to perform an exeresis of the degenerated tendon. After the operation, the patient is directed to the recovery room where the responsible doctor will perform a physical examination and examination before leaving the center.
  This process will take place at the major ambulatory surgery center of the investigator's hospital.
  Arms: Cytokine rich serum injection

SUMMARY:
This study aims to compare arthroscopic resection (surgical intervention) versus infiltration of cytokine rich serum (CRS) (proteins derived from the patient's own blood) for the treatment of lateral epicondylitis (LE).

DETAILED DESCRIPTION:
Lateral epicondylitis (LE) is a common debilitating condition that affects the extensor muscles of the forearm at its junction with the lateral humeral epicondyle. This pathology is commonly treated by a surgical intervention. However, advances in research have allowed the discovery of new and less invasive techniques for its treatment, for example the infiltration of cytokine rich serum.

The aim of the study is to compare the common treatment of this pathology, arthroscopic resection (surgical intervention) with a new technique, infiltration of cytokine rich serum (CRS) (proteins derived from the patient's own blood) with respect to medium and long-term pain reduction.

The study will include a total of 86 patients. Patients will be included by randomization into two groups:

* GROUP 1: 43 patients will be treated with 2 infiltrations of cytokine rich serum.
* GROUP 2: 43 patients will be treated by a regular surgical treatment consisting of arthroscopic resection.

The main objective of this study is to evaluate the efficacy of CRS as compared to arthroscopic resection in reducing pain in the medium term (6 months) in patients with chronic lateral epicondylitis.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Patients with persistent pain (EVA > 5) at lateral epicondyle level of at least 3 months duration.
* Patients with a diagnosis of chronic lateral epicondylitis confirmed with a complementary diagnostic test such as Echo or MRI.
* Availability to follow the study protocol for up to 24 months.
* Patients with the ability to understand study information and give informed consent.
* Patients who sign informed consent.
* Normal hematologic parameters.

Exclusion Criteria:

* Local infection present.
* Patients who have been treated with corticosteroid infiltrations in the same area in the past 4 months.
* Patients who have received treatment with growth factors, PRP, cytokines, or new drug treatments in the same area in the last 12 months.
* Pregnancy or breast-feeding.
* Neoplastic disease.
* Patients being treated with immunosuppressants (medical evaluation).
* Patients undergoing arthroscopic surgery of the same elbow.
* Active liver disease.
* Immunosuppressive or immunodeficiency states.
* Coagulation deficit or abnormalities.
* Thrombocytopenia.
* Treatment with anticoagulants.
* Difficulty understanding and following study procedures.
* Participation in a clinical trial with medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain assessment | 6 months
  reduction of pain to 6 months measured with the Visual Analogue Scale (EVA) scale. The specification of the efficacy parameter is an absolute improvement of the 2-point scale.

SECONDARY OUTCOMES:
Pain assessment with Visual Analogue Scale (EVA) scale | 15 days, 1-3-12-24 months after intervention
  Visual Analogue Scale (EVA) from 0 to 10 points, being 0 no pain, and 10 maximum pain
Patient-Related Tennis Elbow Evaluation (PRTEE) | 15 days, 1-3-6-12-24 months after intervention
  The Patient-Rated Tennis Elbow Evaluation questionnaire (PRTEE) is a specific questionnaire available for assessing the health status of patients with lateral epicondylitis. It is a is a 15-item questionnaire allows patients to rate their levels of tennis elbow pain and disability from 0 to 10, and consists in two subscales:
  1. PAIN subscale (0 = no pain, 10 = worst imaginable) - 5 items
  2. FUNCTION subscale (0 = no difficulty, 10 = unable to do) Specific activities - 6 items Usual activities - 4 items
Grip force | 15 days, 1-3-6-12-24 months after intervention
  measured with a palm grip dynamometer, in kilos
occurrence of pain with resisted wrist extension | 15 days, 1-3-6-12-24 months after intervention
  assessed during medical examination
Number of participants with complications related to the treatment | 15 days, 1-3-6-12-24 months after intervention
  assessed during medical examination
Revision of anti-inflammatory medication and its dose | 15 days, 1-3-6-12-24 months after intervention
  assessed during medical examination

CONTACTS AND LOCATIONS:
Overall Officials: Mònica Salomó, MD, Principal Investigator — Corporacion Parc Tauli
Locations (2):
- Spain (2):
  - Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No